CLINICAL TRIAL: NCT06499857
Title: Semaglutide for Metabolic Intervention and Adipose Loss to Treat Atrial Fibrillation
Acronym: SEMINAL-AF
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB23-0889
Record Dates: First submitted 2024-04-24; First posted 2024-07-15 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Overweight or Obesity; Atrial Fibrillation
MeSH Terms: conditions — Overweight; Obesity; Atrial Fibrillation | interventions — semaglutide

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Prospective, Randomized and Blinded
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Semaglutide (Active Comparator): Participants will have a 2 in 3 chance of receiving semaglutide (2.4 mg).
  Interventions: Drug: Semaglutide
- Placebo (Placebo Comparator): Participants will have a 1 in 3 chance of receiving placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Semaglutide — 3ml pen-injector containing semaglutide 3.0mg/ml solution for subcutaneous use.
  Arms: Semaglutide
Drug: Placebo — 3ml pen-injector containing placebo solution for subcutaneous use.
  Arms: Placebo

SUMMARY:
The goal of the study is to learn how a weight loss medication called semaglutide, which is used to treat obesity, in addition to standard AF treatment might affect AF, atrial fibrillation severity, and whether it changes the risk of atrial fibrillation recurring after standard AF treatments.

DETAILED DESCRIPTION:
Obesity and atrial fibrillation (AF) pose a significant burden on healthcare systems worldwide. Obesity is an established independent risk factor for both the development of AF, as well as increased disease severity and adverse outcomes. According to a meta-analysis of 51 studies involving 60,000 individuals, every 5-unit increment in BMI confers an additional 19%-29% risk of incident AF, a 10% risk of post-operative AF, and a 13% risk of post-ablation AF. The estimated prevalence of AF in the United States is approximately 5.2 million, and is expected to increase to 12.1 million by the year 2030, likely explained by mirroring the growth of the obesity epidemic. While many associations have been made, the underlying pathophysiological mechanisms linking obesity and AF are incompletely understood.

Two large longitudinal cohort studies demonstrated that obesity contributes to disease progression to persistent or permanent forms of AF. Importantly, significant weight loss achieved by bariatric surgery has been associated with a reduction in the risk of new-onset AF by 29% in the prospective matched cohort Swedish Obese Study. Weight loss achieved with intensive lifestyle modification has also been shown to impact AF burden. However, these studies have not systematically investigated the biological mechanisms underlying weight loss and AF.

The novelty of the proposed study is that it will be the first to examine the impact of weight loss with semaglutide 2.4 mg on biological signaling and cardiac remodeling in relation to reductions in AF burden. Additionally, the proposed study will be the first to evaluate the effect of pharmacological weight loss on the risk of arrhythmia recurrence, combined with antiarrhythmic drugs (AAD) and/or catheter ablation (CA), which are the current first-line strategies for rhythm maintenance in patients with obesity. That is relevant as obesity is a chronic and relapsing health condition as demonstrated in multiple large intensive lifestyle modification studies which show a significant weight loss in the short term but minimal weight reduction in the long-term follow up. Pharmacotherapy has been shown to be superior to lifestyle modification to achieve larger and maintained weight loss.

Therefore, The investigators propose the first-ever double-blinded placebo controlled randomized clinical study to assess the efficacy and impact of an anti-obesity medication on atrial fibrillation in patients receiving contemporary therapies for atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years
2. BMI greater than or equal to 30 kg/m2
3. Paroxysmal AF or persistent AF, in whom catheter ablation (CA) for AF is expected within 1 year (A group) or in whom catheter ablation is NOT expected within 1 year (M group)
4. Ability to provide informed consent before any trial-related activities.
5. Patients with type 2 diabetes mellitus (T2DM) will be included:

   1. If HbA1c (glycated hemoglobin) is less than or equal to 10 %
   2. If the subject is taking basal insulin only or oral hypoglycemic agents or a combination of those.
   3. Patients on SGLT2-inhibitors and TZDs (Thiazolidinedione) will be included if they have been on a stable dose of these medications for at least 6 months
   4. The following protocol will be adopted to adjust insulin secretagogues (sulfonylureas or meglitinides) and insulin during the study (adapted from the Look Ahead Study).

Patients will be asked to check their blood glucose (BG) 4 x day (before meals and at bed time) during the dose escalation and dose stabilization phases (weeks 0 to 20) and recommendation of dose adjustments will be immediately sent to their treating physician according to the dose adjustment scale below:

* 2 blood sugars <100 mg/dl- reduce meds [insulin secretagogues (sulfonylureas or meglitinides) and basal insulin] by 0-50 %
* 3 blood sugars 80-100 mg/dl- reduce meds [insulin secretagogues (sulfonylureas or meglitinides) and basal insulin] by 25-75%
* 3 blood sugars <80 mg/dl > 2 x week or severe hypoglycemia or symptomatic hypoglycemia- reduce meds [insulin secretagogues (sulfonylureas or meglitinides) and basal insulin] by 50-100 %

Randomization to treatment (active and placebo) will be stratified to balance patients with T2DM across the study arms. After completion of the trial a prespecified subgroup analysis of the patients enrolled affected by T2DM will be performed.

For women of child-bearing potential, use of appropriate contraception will be required.

In patients that are prescribed amiodarone, standard care practices will be implemented to evaluate for liver and thyroid side effects with baseline liver and thyroid function tests via blood draw and evaluation every 6 months.

Exclusion Criteria:

1. Current use of GLP-1 RA (glucagon-like peptide receptor agonists) or DPP4 (Dipeptidyl peptidase-4)-inhibitors or use within the last 90 days prior to screening
2. Current antiobesity medication use or use within the last 90 days prior to screening
3. A self-reported change in body weight of > 5 kg (11 lb.) within 30 days before screening
4. History of bariatric surgery
5. History of type I diabetes mellitus
6. Current use of prandial insulin
7. Hospitalization for unstable angina, or TIA (Transient ischemic attack) < 30 days prior to screening
8. Pulmonary embolism < 90 days before screening
9. MI (myocardial infarction), stroke, etc. < 90 months prior to screening
10. Uncontrolled thyroid disease: TSH (Thyroid-stimulating hormone) > 10.0 mIU/L (Milli-international Units Per Liter) or < 0.4 mIU/L (Milli-international Units Per Liter) at screening
11. Active malignancy
12. Active enrollment in another investigational study that includes any kind of intervention
13. The receipt of any investigational drug within 90 days prior to this trial.
14. Inability to comply with study procedures
15. Acute pancreatitis < 180 days before screening
16. History or presence of chronic pancreatitis
17. CKD (Chronic Kidney Disease) stage 4 (GFR <30 ml/min)
18. A personal or family history of medullary thyroid carcinoma (MTC) or Multiple Endocrine Neoplasia syndrome type 2 (MEN 2)
19. A prior serious hypersensitivity reaction to semaglutide or to any of the excipients in WEGOVY
20. Chronic inflammatory conditions requiring immunosuppression and/or on glucocorticoids
21. Previous participation in this trial (received at least one dose of study drug or placebo)
22. Pregnant, breast-feeding or planning pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Time to first AF event detected by routine outpatient monitoring | Baseline to Week 68
  Defined by length of time detected by routine outpatient monitoring (Holter, mobile telemetry, or implantable loop recorder).
Change from baseline in AF burden detected by routine outpatient monitoring. | Baseline to Week 68
  Defined as the percentage of time spent in atrial fibrillation as detected by routine outpatient monitoring (Holter, mobile telemetry, or implantable loop recorder).

SECONDARY OUTCOMES:
Weight loss | Baseline to Week 68
  Change in Weight (kilograms) measured.
Change in waist circumference | Baseline to Week 68
  Change waist circumference (cm) measured.
Change in epicardial and/or pericardial adipose tissue volume | Baseline to Week 68
  Decrease measured by Cardiovascular magnetic resonance
Change in left and right ventricular size (mass) | Baseline to Week 68
  Change in left and right ventricular size derived from time volume curves, and left and right atrial volumes (mL) measured by cardiovascular magnetic resonance
Change in left and right ventricular size (volume) | Baseline to Week 68
  Change in left and right ventricular size derived from time volume curves, and left and right atrial volumes (mL) measured by cardiovascular magnetic resonance
Change in left and right ventricular function (ejection fraction) | Baseline to Week 68
  Change in left and right ventricular function derived from time volume curves, and left and right atrial volumes (mL) measured by cardiovascular magnetic resonance
Change in left ventricular strain | Baseline to Week 68
  Change in left ventricular strain derived from time volume curves, and left and right atrial volumes (mL) measured by cardiovascular magnetic resonance
Change in left ventricular diastolic parameters | Baseline to Week 68
  Change in left ventricular strain diastolic parameters measured by cardiovascular magnetic resonance
Change in LV (left ventricular) myocardial fibrosis | Baseline to Week 68
  Decrease in LV (%)myocardial fibrosis burden as measured by changes in native myocardial T1 times (milliseconds) measured by Cardiovascular magnetic resonance
Change in sympathetic activity and in circulating cytokines and adipokines | Baseline to Week 68
  Decrease in systemic inflammation as measured by the levels of circulating cytokines and adipokines such as [CRP(C-reactive protein), TNF(Tumor necrosis factor), IL-6 (Interleukin 6), IL-1 alpha beta IL-8, IL-10, 16-18 monocyte chemoattractant protein (MCP-1), VEGF (Vascular endothelial growth factor)] (pg/mL) and adipokines (leptin, adiponectin, resistin, and visfatin) (pg/mL).
Change in Autonomic tone as determined by heart rate variability | Baseline to Week 68
  HRV (milliseconds) will measured from baseline to Week 68 by outpatient rhythm monitoring
Changes from baseline through Week 68 of Atrial conduction times | Baseline to Week 68
  Estimated by simple P wave duration (milliseconds) measured by 12-lead ECG
Changes in Body mass composition | Baseline to Week 68
  Change in Body mass composition (percentage) measured by bio-impedance
Changes in Metabolic effects | Baseline to Week 68
  Metabolic effects measured by CMP/HgA1C (mg/dL and %)
Left atrial and myocardial stress | Baseline to Week 68
  Change measured by Serum BNP (pg/mL), which reflects left atrial and myocardial stress
Changes from baseline through Week 68 of novel Patient Reported Outcome Assessment. | Baseline to Week 68
  Detection of within-patient changes on impact of health on an individual's everyday life reported in a novel Patient-Reported Outcome Assessment between baseline and Week 68.

CONTACTS AND LOCATIONS:
Overall Officials: Silvana Pannain, MD, Principal Investigator — University of Chicago
Locations (2):
- United States (2):
  - The University of Arizona College of Medicine- Phoenix, Phoenix, Arizona
  - University of Chicago, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No